CLINICAL TRIAL: NCT04923425
Title: Gustatory Modulators Among a Sample of Depressed Egyptian Adults Under Anti-depressants Therapy. A Retrospective Cohort Study
Brief Title: Gustatory Modulators Among a Sample of Depressed Egyptian Adults Under Anti-depressants Therapy
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Christine Raouf George Mikhail, Principal Investigator, Cairo University
Other Study IDs: 18936 CairoU
Record Dates: First submitted 2021-06-06; First posted 2021-06-11 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Taste Disorders
MeSH Terms: conditions — Taste Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Exposure 1: commonly prescribed tricyclic antidepressants (Imipramine, Amitriptyline, Clomipramine HCL) administered for at least 3 months
- Exposure 2: commonly prescribed Selective Serotonin Re-uptake inhibitors antidepressants ( Fluoxetine, Fluvoxamine, Sertraline, Citalopram, Paroxetine) administered for at least 3 months
- Non exposure: Non-pharmacological treatment (psychotherapy)

SUMMARY:
Identify possible modulators for developing gustatory dysfunction among a sample of depressed Egyptian adults (age from 20 to 50 years old) under anti-depressants therapy ( for at least 3 months) using a questionnaire ( appendix) with a binary measuring unit (yes/no).

DETAILED DESCRIPTION:
PECO

* P Population: depressed Egyptian adults under anti-depressants therapy
* E1 Exposure 1: commonly prescribed tricyclic antidepressants (Imipramine, Amitriptyline, Clomipramine HCL)
* E2 Exposure 2: commonly prescribed Selective Serotonin Re-uptake inhibitors antidepressants ( Fluoxetine, Fluvoxamine, Sertraline, Citalopram, Paroxetine)
* C control (non exposure) : non-pharmacological treatment ( psychotherapy)
* O Outcome: Identify possible gustatory dysfunction modulators among these patients using a questionnaire ( appendix) with a binary measuring unit (yes/no).

ELIGIBILITY:
Inclusion Criteria:

* • Depressed Egyptian adults under antidepressants therapy for at least 3 months/non-pharmacological treatment( psychotherapy)

  * Age from 20 to 50 years old

Exclusion Criteria:

* Antipsychotics

  * Hypnotics
  * Anticonvulsants
  * Ages other than the mentioned • Olfactory dysfunction
  * Chemosensory dysfunction

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Depressed Egyptian adults under anti-depressants therapy The patients will be recalled using their phone numbers recorded in their follow up records in order to come to the Diagnosis center at the faculty of Dentistry, Cairo University to be assessed for possible gustatory dysfunction modulators and will be given identification numbers and divided into three groups, to which the operator shall be blinded.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-02-22 (Actual); Primary Completion 2020-08-08 (Actual); Study Completion 2020-10-07 (Actual)

PRIMARY OUTCOMES:
Gustatory dysfunction modulators | during a period of 7months from February 2020 till August 2020
  -C.M will use an assessment questionnaire (appendix) to assess possible modulators for developing gustatory dysfunction including a number of short-term and long-term factors such as body mass, gender, age, local and systemic diseases, excessive alcohol drinking, drug dependence, smoking, state of oral hygiene, consumption of some foods or drugs

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No